CLINICAL TRIAL: NCT07317713
Title: A Two-decade Mortality Risk Analysis of Gastrointestinal Carcinoid Neoplasms: an Updated SEER-based Study 2000-2022
Status: Completed | Type: Observational
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, asmaa salama ibrahim, Resident physician of gastroenterology, Suez Canal University
Other Study IDs: A277
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Carcinoid Tumor
MeSH Terms: conditions — Carcinoid Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Carcinoid tumors are rare neuroendocrine tumors with slowly progressive course with the sites are small intestine accounting for 45%, rectum (20%), appendix (17%), colon (11%), and stomach (7%). This study focus on the mortality risk analysis for GI carcinoids due to data insufficiency in the literature.

DETAILED DESCRIPTION:
Carcinoid tumors are rare neuroendocrine tumors with slowly progressive course with the sites are small intestine accounting for 45%, rectum (20%), appendix (17%), colon (11%), and stomach (7%). This study focus on the mortality risk analysis for GI carcinoids due to data insufficiency in the literature. This is a retrospective cohort study based on the Surveillance, Epidemiology, and End Results (SEER) database using SEER*Stat software covering approximately 28% of the U.S. The inclusion criteria involved all patients with primary malignant GI carcinoid tumor diagnosed between 2000 and 2021 with sequence number 0 or 1. Sequence 0 indicated the patient had only one cancer record while sequence 1 indicated the patient may had developed many cancer records following the first one. In addition, the tumors were restricted to malignant behavior codes (ICD-O-3 Code 3). We used SEER*Stat software (version 9.0.42.0) to conduct data extraction and statistical analysis. We used the MP-SIR session to calculate the SMR as Observed/Expected (O/E) with a 95% confidence interval (CI) and the excess risk (ER) was per 10,000. Statistical significance was achieved at 0.05. With further analysis, we compared cancer as a cause of death (COD) to other non-cancer COD across different time intervals and primary sites among GI carcinoid tumour.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with gastrointestinal carcinoid tumor
* from 2000-2022
* histologically confirmed

Exclusion Criteria:

* death certificate only and autopsy only patients
* patients with unknown age data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The inclusion criteria involved all patients with primary malignant GI carcinoid tumor diagnosed between 2000 and 2022 with sequence number 0 or 1. Sequence 0 indicated the patient had only one cancer record while sequence 1 indicated the patient may had developed many cancer records following the first one. In addition, the tumors were restricted to malignant behavior codes (ICD-O-3 Code 3).
Sampling Method: Non-Probability Sample
Enrollment: 93481 (Actual)
Dates: Start 2000-12-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
The standardized mortality ratio of GI carcinoid tumors | 2000-2022
  SEER*Stat software (version 9.0.42.0) was used to conduct data extraction and statistical analysis. The MP-SIR session was used to calculate the SMR as Observed/Expected (O/E) with a 95% confidence interval (CI) and the excess risk was per 10,000. Statistical significance was achieved at 0.05. With further analysis, we compared cancer as a cause of death to other non-cancer causes of death across different time intervals and primary sites among GI carcinoid tumour.

IPD SHARING:
Plan to Share IPD: Undecided